CLINICAL TRIAL: NCT00790504
Title: Prospective Follow up of the Female Pelvic Floor in Multiple Gestation Using Transperineal Ultrasound
Brief Title: Transperineal Ultrasound for the Female Pelvic Floor in Women With Multiple Gestation
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty recruiting patient. Lack of research assistant.
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Vered Eisenberg, MD, Sheba Medical Center
Other Study IDs: SHEBA-08-5470-VE-CTIL
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Pregnancy
Keywords: Pelvic floor; Transperineal ultrasound; Multiple pregnancy; Singleton pregnancy; Female pelvic floor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 study group: Women with multiple gestations recruited from the prenatal care or high risk pregnancy units
- 2 control group: Women with singleton gestation recruited from the prenatal care or high risk pregnancy units

SUMMARY:
This trial studies the effect of pregnancies of multiple gestations (i.e. twins, triplets etc.) on the female pelvic floor with regards to the pregnancy itself and labor and delivery mode, by using transperineal ultrasound. This will be compared with pregnancies with single fetuses.

DETAILED DESCRIPTION:
This trial studies the effect of pregnancies of multiple gestations (i.e. twins, triplets etc.) on the female pelvic floor with regards to the pregnancy itself and labor and delivery mode, by using transperineal ultrasound. This will be compared with pregnancies with single fetuses. See study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women with multiple gestations
* Women with singleton gestation
* Able to understand the consent form

Exclusion Criteria:

* None specified

Ages: 17 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with multiple gestations recruited from the prenatal care or high risk pregnancy units
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Multiple gestation affects the pelvic floor more than singleton gestation | Until recruitment completion

SECONDARY OUTCOMES:
The mode of delivery affects pelvic floor outcome | As above

CONTACTS AND LOCATIONS:
Overall Officials: Vered H Eisenberg, MD MHA, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel